CLINICAL TRIAL: NCT03715257
Title: Evaluation of Advanced Extubation Techniques in Bariatric Surgery: A Randomized Controlled Prospective Study
Brief Title: Evaluation of Advanced Extubation Techniques in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, EMİNE YURT, clinical researcher, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: KIA 2018/19
Record Dates: First submitted 2018-07-27; First posted 2018-10-23 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Bariatric Surgery Candidate; Extubation
Keywords: Advanced extubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14F staged extubation set guidewire (Active Comparator): 14F staged extubation set guidewire is a single use supraglottic airway device. This airway device provides access and functional separation of the respiratory and digestive tracts.
  Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are recorded for the first 20 postoperative minutes. Blood gas analyses are done before extubation and 15 minutes after placement of the extubation catheter.
  The patients are randomly distributed into two groups; one with 14F staged extubation set guidewire (n=50)
  Interventions: Device: 14F staged extubation set guidewire
- Tube changing catheter (Active Comparator): Tube changing catheter is an alternative extubation device. Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are recorded for the first 20 postoperative minutes. Blood gas analyses are done before extubation and 15 minutes after placement of the extubation catheter.
  The patients are randomly distributed into two groups; one with 14F staged extubation set guidewire (n=50)
  Interventions: Device: Tube changing catheter

INTERVENTIONS:
Device: 14F staged extubation set guidewire — 14F staged extubation set guidewire is a single use supraglottic airway device. This airway device provides access and functional separation of the respiratory and digestive tracts.
  Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are recorded for the first 20 postoperative minutes. Blood gas analyses are done before extubation and 15 minutes after placement of the extubation catheter.
  The patients are randomly distributed into two groups; one with 14F staged extubation set guidewire (n=50)
  Arms: 14F staged extubation set guidewire
Device: Tube changing catheter — Tube changing catheter Tube changing catheter is an alternative extubation device. Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are recorded for the first 20 postoperative minutes. Blood gas analyses are done before extubation and 15 minutes after placement of the extubation catheter.
  The patients are randomly distributed into two groups; one with 14F staged extubation set guidewire (n=50)
  Arms: Tube changing catheter

SUMMARY:
The aim of prospective clinic study is to compare the tolerance and effectivity of Cook tube changing catheter and staged extubation set following laparoscopic morbid obesity surgery. The use of step extubation in difficult extubation is life-saving. The use of cascade extubation set in morbid obese and especially bariatric surgery patients is also life-saving.

DETAILED DESCRIPTION:
Extubation in difficult airway can be defined as transition from a controlled environment to an uncontrolled. According to the results of the NAP4 study conducted in England, one third of the anaesthesia related major airway complications occur during awakening or compilation and the mortality rate was 5%. The Difficult Airway Society extubation guideline published in 2015 suggested awake extubation in patients with risk for airway or systemic risk factors, and mentioned about the importance of the benefit from further techniques such as Bailey maneuver, remifentanyl technique and tube changing catheters. The aim of prospective clinic study is to compare the tolerance and effectivity of Cook tube changing catheter and staged extubation set following laparoscopic morbid obesity surgery.

The Cook staged extubation set (Cook Medical) has been developed to facilitate management of the difﬁcult airway. A guidewire inserted before tracheal extubation provides access to the subglottic airway should re-intubation be required. This prospective study examines patients' tolerance of the guidewire and its impact on clinical status around tracheal extubation in the postoperative unit.Vital signs, incidence of symptoms and patient tolerance of the wire are recorded.

MATERIAL AND METHOD

Researches conduct a prospective study using the Cook staged extubation set in 100 patients undergoing tracheal extubation in the operation room of Derince hospital.

Local ethics committee approval and written informed consent are planned to work with 100 patients.The patients are randomly distributed into two groups; one with 14F staged extubation set guidewire (n=50)and the other with tube changing catheter (n=50). Cuff leakage test is done prior to extubation and 3 mg/kg intravenous sugammadex is administered. The patients who reached the awake extubation criteria are extubated using one of the above catheters. Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are recorded for the first 20 postoperative minutes. Blood gas analyses are done before extubation and 15 minutes after placement of the extubation catheter.

During the procedure, the patient's blood pressure, heart rate, oxygen saturation, any complications that may develop will be recorded.

Induction of anesthesia; difficult airway management, difficult mask and / or difficult intubation incidence, Mallampati scores, the use of one of the difficult intubation techniques during intubation (such as FastTrack, videolaryngoscopy or fiberoptic intubation), perioperative mechanical ventilation parameters (ventilation mode, tidal volume, respiratory frequency, end of tidal CO2 (carbon dioxide) pressure, PEEP usage, SpO2 (saturation oxygen), airway peak pressure, urine volume, arterial blood gas parameters are recorded.Patients receive intravenous lidocaine at a dose of 1 mg / kg before induction and extubation. Prednisolone 1 mg / kg intravenous is given when necessary, such as laryngospasm development or recurrent airway manipulations. Duration of operation, surgical method (laparotomy / laparoscopy), agents used in induction and postoperative analgesia, use of blood, blood product and vasopressor are recorded. Before extubation, the cuff leakage test is performed and the extubations are made at a height of 30-35º degree. In the induction and maintenance of anesthesia, patients are given propofol 2 mg / kg, rocuronium 0.6 mg / kg, fentanyl 1mcg / kg and sevoflurane 2%. For extubation sugammadex is given iv at a dose of 3 mg / kg.

In patients who were extubation with cook staged extubation set; coughing, straining, hemodynamic parameter change, 20% heart rate and / or changes in arterial blood pressure and presence of hypoxemia (SpO2 <94%) are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Patients who have undergone obesity surgery
* ASA 2-3 patients
* Patients who have received written informed consent

Exclusion Criteria:

* Patients under the age of 18
* Patients refusing to participate in the study
* Patients under emergency conditions
* Earlier laryngeal and tracheal surgery, those who undergo lung surgery
* Those with allergies to lidocaine
* Patients with FEV1 / FVC below 60%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
obese patient's cook staged extubation set tolerance (guidewire and tube changing catheter) | Up to 20 minutes (after extubation at minute 0, 5,10,15,20)
  In patients who were extubation with cook staged extubation set; coughing, straining, hemodynamic parameter change, 20% heart rate and / or changes in arterial blood pressure and presence of hypoxemia (SpO2 <94%)

SECONDARY OUTCOMES:
Successful tracheal extubation and 14F staged extubation set guidewire patient tolerance | Up to 20 minutes (after extubation at minute 0, 5,10,15,20)
  Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are records for the first 20 postoperative minutes.
Successful tracheal extubation and tube changing catheter patient tolerance | Up to 20 minutes (after extubation at minute 0, 5,10,15,20)
  Tolerance of the patient to the catheter coughing, straining reflex. Cough, straining, hemodynamic parameters and occurrance of hypoxemia (SpO2<94%) are records for the first 20 postoperative minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Yurt, Study Director — Anesthesiology
Locations (1):
- Kocaeli Derince Education and Research Hospital, Derince, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No